CLINICAL TRIAL: NCT05378828
Title: Interest of Using an Electric Wheelchair Equipped With Anti-collision Sensors to Improve the Driving Confidence of Elderly People in EHPAD
Brief Title: Interest of Using an Electric Wheelchair Equipped With Anti-collision Sensors for Elderly People in EHPAD
Acronym: SWADAPT4
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties encountered that were not highlighted in previous studies (traffic situations that made daily life difficult for users, need to rework the system)
Sponsor: Pôle Saint Hélier (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other); Centre Communal d'Action Sociale Saint-Etienne (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-A03138-33
Record Dates: First submitted 2022-05-05; First posted 2022-05-18 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of an electric wheelchair with or without sensors (Other): During 3 weeks, the electric weehlchair will not have sensors, then sensors will be put on the wheelchair for the next 3 weeks then removed for 3 other weeks.
  Interventions: Device: Using anti-collision Sensors on electric wheelchairs; Other: Use of an electric wheelchair without sensors

INTERVENTIONS:
Device: Using anti-collision Sensors on electric wheelchairs — use of anti-collision sensors on the electric wheelchair during 3 weeks
Other: Use of an electric wheelchair without sensors — Use of an electric wheelchair without sensors for 3 weeks before using anti-collision sensors then during 3 weeks after using the anti-collision sensors.

SUMMARY:
The device which is the subject of this investigation is a robotic assistance module for the driving of a semi-autonomous electric wheelchair (FRE). It's intended to accessorize the FRE to improve the safety conditions during the driving of a FRE, making it possible to decrease the rate of accident in wheelchair on the one hand, increase the confidence of driving on the other hand, and facilitate the access to the FRE of people not being able to aspire to it without the use of a device of safety of this type.

ELIGIBILITY:
Inclusion Criteria:

* Over 60 years of age,
* Resident in an institution for the elderly or nursing home,
* with a electric wheelchair but expressing driving difficulties
* Having freely consented to participate in the study,
* In the case of a guardianship, the legal representative having read the information document intended for the legal guardian of an adult under legal protection (under guardianship) and having given his or her free and informed consent for the person for whom he or she is responsible to participate in the study (in agreement with the patient).

Exclusion Criteria:

* Impaired comprehension preventing the protocol from being carried out,
* Person in an emergency situation unable to give prior consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Evaluate benefits of using a FRE equipped with the assistance module on the confidence in driving electric wheelchair for elderly people in EHPAD | Day 42
  Evaluation by using the under score of confidence of Wheelchair Skill Test questionnaire (WST-Q-T 5.1) during the period of use of the module and at the end.
  The score goes from 0 to 56 (56 is the higher level of confidence).

SECONDARY OUTCOMES:
Driving habilities | Day 42 and Day 63
  Benefits of the sensors on ability and performance of tasks performed with the electric wheelchair by Wheelchair Skill Test questionnaire (WST-Q-T 5.1).
  The score will go from 0 to 56 for each scale (performance and frequency), a high score will represent a good driving performance
Distance traveled measured by sensors on the FRE | Day 21, Day 42 and Day 63
  The distance will be measured in meters with a lap counter type.
Mesure of mental load related to wheelchair mobility | Day 21, Day 42 and Day 63
  Mental load will be measured by the NASA-Task Load Index. It is in the form of six scales where the participant must assign a score between zero and one hundred to each of them, score indicating a growing level of intensity. Three dimensions relate to the demands imposed on the subject (mental, physical and temporal demands) and three to the interaction of a subject with the task (effort, frustration and performance).
Ease of Use Questionnaire | Day 42
  Satisfaction of using FRE by users will be mesured by the Ease of Use Questionnaire. He is composed of 27 questions, each question is valued between 0 to 7. a high score will represent a high satisfaction.
Acceptability of anti-collision sensors by users | Day 42
  A acceptability questionnaire based on the Unified Theory of Acceptance and Use of Technology (UTAUT) will be completed at day 42, with semi-directive interview

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Pôle Saint-Hélier, Rennes, Brittany Region
  - CCAS Saint-Etienne, Saint-Etienne
  - USLD Saint Etienne, Saint-Etienne